CLINICAL TRIAL: NCT01882985
Title: A Phase II Study to Evaluate the Effects of Docetaxel Plus Lycopene in Castration Resistant, Chemotherapy-Naïve Prostate Cancer Patients
Brief Title: Docetaxel Plus Lycopene in Castration Resistant, Chemotherapy-Naïve Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, John P. Fruehauf, Professor of Clinical Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 10-11 [HS# 2010-7765]; 2010-7765 (Other: University of Calfornia, Irvine); NCI-2011-00037 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
Keywords: docetaxel; lycopene; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Lycopene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (docetaxel and lycopene) (Experimental): Patients receive docetaxel IV over 1 hour on day 2 and lycopene PO once daily on days 1-21. Treatment repeats every 21days for at least 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Dietary Supplement: Lycopene

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: 114977-28-5; 40466; 628503; RP 56976; RP56976; Taxotere; TXT
Dietary Supplement: Lycopene — Given PO
  Other Names: 407322; 502-65-8; all-trans-Lycopene; Lyc-O-Mato; LYCO; psi; psi-Carotene

SUMMARY:
This phase II trial evaluated the impact of giving docetaxel together with lycopene supplements in treating patients with hormone-resistant prostate cancer not previously treated with chemotherapy. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemoprevention is the use of certain drugs, such as lycopene, to keep cancer from forming. Giving docetaxel together with lycopene may be an effective treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the prostate-specific antigen (PSA) response rate according to the criteria of Bubley, et al. (>50% reduction from baseline) in subjects treated with a combination of docetaxel and lycopene.

SECONDARY OBJECTIVES:

I.To determine the objective response rate (ORR) according to modified RECIST criteria in patients with measurable disease, following treatment with docetaxel and lycopene.

II. To define the time to PSA progression, according to the response criteria of Scher, et al., in subjects treated with docetaxel and lycopene.

III. To determine the safety and tolerability of lycopene in combination with docetaxel.

IV. To determine the effects of docetaxel + lycopene therapy on the functioning of the IGFR-I, selected biomarkers, and docetaxel blood levels in plasma and peripheral blood mononuclear cells (correlative studies).

OUTLINE:

Patients receive 75 mg/m2 docetaxel intravenously (IV) over 1 hour q 21 days and lycopene 30 mg capsules orally (PO) once daily on days 1-21. Treatment repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histological diagnosis of adenocarcinoma of the prostate and 2 rising pre-study PSA values >= 1 ng/ml at least 1 week apart within 28 days prior to enrollment
* Patients must be unresponsive to androgen-deprivation therapy (ADT), as indicated by a rising PSA level above the ADT nadir
* Patient must not have received chemotherapy, biologic therapy, or any other investigational drug for any reason within 28 days prior to start of therapy, and must have recovered from toxicities of prior therapy to grade 1 or less
* Patients must have been surgically or medically castrated; if the patient is being treated with medical castration, he must be willing to continue this treatment for the duration of the study; ADT should not be initiated, terminated, or dose-adjusted during the study
* Prior external beam radiation therapy (to less than 30% of the bone marrow only) is allowed; at least 28 days must have elapsed since the completion of radiation therapy and the patient must have recovered from side effects; prior treatment with samarium-153 or strontium-86 is allowed if at least eight weeks have elapsed since dosing, and all toxicities have resolved to grade 1; soft tissue disease which has been radiated in the prior 2 months is not assessable as measurable disease
* Patients may have received prior surgery; however, at least 21 days must have elapsed since completion of surgery and the patient must have recovered from all side effects
* Normal serum bilirubin and serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvate transaminase (SGPT) =< 1.5 x the institutional upper limit of normal obtained within 14 days prior to start of therapy; liver function tests should be evaluated prior to each treatment
* Serum creatinine =< 1.5 x the institutional upper limit of normal obtained within 14 days prior to start of therapy
* Men of child bearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count >= 1,500/microliter (mcL)
* Hemoglobin of >= 8.0gm/dL
* White blood cell count > 2,500/mcL
* Platelets >= 100,000/mcL
* Patients with lower values may participate if, in the opinion of the investigator, the cytopenias are the result of bone marrow involvement with active prostate cancer
* Patients must be able to take oral medications
* All patients must be informed and must sign and give written informed consent in accordance with institutional and federal guidelines; patients who are unable to comply with study and/or follow-up procedures are ineligible

Exclusion Criteria:

* Uncontrolled brain or spinal cord metastases
* History of congestive heart failure or myocardial infarction within the previous six months
* History of allergy or hypersensitivity to any component of the study drugs
* Evidence or history of a bleeding diathesis or coagulopathy, including therapy-induced coagulopathy
* Presence of chronic diarrhea (> grade 1 by Common Toxicity Criteria (CTC)), short bowel syndrome, pancreatic insufficiency, or malabsorption
* Presence of any severe or uncontrolled concurrent medical condition which, in the opinion of the investigator, would increase the risk of serious toxicity from the study drugs
* Concurrent use of any vitamin, herb, or mineral supplements for at least 14 days prior to start of therapy

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Fruehauf, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Docetaxel and Lycopene)
Started | 14
Completed | 12
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Docetaxel and Lycopene)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Proporation of Subjects Achieving Partial Response, Stable Disease or Progressive Disease Based on PSA Response Rates
Description: To define the prostate-specific antigen (PSA) response rate according to the criteria of Bubley, et al. in subjects treated with a combination of docetaxel and lycopene. Per criteria of Bubley, et al., PSA response rate is defined the number of subjects who achieve a >50% decline in PSA from baseline.
Time Frame: Up to week 12 of therapy
Population: One patient was inevaluable due to lost to follow up and one patient withdrew consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Docetaxel and Lycopene)
Number analyzed (Participants) | 12
Participants
  Partial Response (PR) | 9
  Stable Disease (SD) | 2
  Progressive Disease (PD) | 1

2. Secondary Outcome: Objective Response Rate as Assessed by RECIST Criteria in Either Visceral or Lymph Node Metastases
Description: The percent of subjects achieving an objective response by RECIST criteria in either visceral or lymph node metastases, and the percent achieving clinical complete disappearance of disease at any site, will be recorded.
Time Frame: Up to 4 years
Population: Data was not collected for this objective.
Arm/Group | Treatment (Docetaxel and Lycopene)
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to PSA Progression
Description: The definition of time to PSA progression is the date (after the initiation of chemotherapy on day 2) that a 25% or greater increase, and an absolute increase of 2ng/mL or more, from the nadir PSA is documented. If there is no decrease in PSA following chemotherapy, then PSA progression is the date for documentation of a 25% increase from the baseline value along with an increase in absolute value of 2ng/mL or more.
Time Frame: Up to 4 years
Population: Mean time to PSA progression
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment (Docetaxel and Lycopene)
Number analyzed (Participants) | 12
days | 335 (350.1)

4. Secondary Outcome: Toxicity of Combined Docetaxel + Lycopene Therapy
Description: The percentage of subjects experiencing grade 3-4 hematologic and non-hematologic toxicity will be recorded, as well as the reason for ending treatment. This outcome measure was not collected due to lack of funding.
Time Frame: Up to 4 years
Population: Data was not collected for this outcome measure.
Arm/Group | Treatment (Docetaxel and Lycopene)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 86 days. Participants can then choose to continue treatment beyond this point until disease progression.
Arm/Group | Treatment (Docetaxel and Lycopene)
All-Cause Mortality (participants affected / at risk) | 2/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Docetaxel and Lycopene) (N=14)
Severe Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac Arrhythmia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Docetaxel and Lycopene) (N=14)
Diarrhea (Gastrointestinal disorders) | 3
Alopecia (Immune system disorders) | 3
Fatigue (General disorders) | 8
Constipation (Gastrointestinal disorders) | 2
Onchomychosis (Skin and subcutaneous tissue disorders) | 5
Insomnia (General disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Edema (Injury, poisoning and procedural complications) | 3
Pain (General disorders) | 3
Anemia (Blood and lymphatic system disorders) | 2
Decreased Appetite (General disorders) | 2
Cracked Tooth (General disorders) | 1
Skin Changes (Skin and subcutaneous tissue disorders) | 1
Left Eye Conjunctivitis (Infections and infestations) | 1
Depression (Psychiatric disorders) | 1
Nausea (General disorders) | 1
Decrease taste (Respiratory, thoracic and mediastinal disorders) | 2
Dry Mouth (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Dehydration (General disorders) | 1
Neuropathy (Nervous system disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Proteinuria (Blood and lymphatic system disorders) | 1
Confusion (General disorders) | 1
Hemorrhoids (Vascular disorders) | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymoses (General disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Blurred Vision (General disorders) | 1
Hot Flashes (General disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Hypertension (Blood and lymphatic system disorders) | 1
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No